CLINICAL TRIAL: NCT04042753
Title: Phase II Trial of Nivolumab Plus Ipilimumab in Patients With Aggressive Pituitary Tumors
Brief Title: Nivolumab and Ipilimumab in People With Aggressive Pituitary Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-216
Record Dates: First submitted 2019-07-31; First posted 2019-08-02 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Pituitary; Pituitary Tumor; Pituitary Carcinoma; Pituitary Cancer
Keywords: Pituitary tumor; Nivolumab; Ipilimumab; 19-216
MeSH Terms: conditions — Pituitary Diseases; Pituitary Neoplasms | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pituitary Cancer (Experimental): Participants will have a pituitary adenoma/carcinoma of any histology
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab 3 mg/kg every 3 weeks,
Drug: Nivolumab — Nivolumab 1 mg/kg every 3 weeks for 4 cycles
Drug: Nivolumab — Following concurrent ipilimumab and nivolumab, patients will receive single agent nivolumab at 480 mg every 4 weeks for 6 cycles (1 cycle=4 weeks) with the option of continuing until disease progression or until the end of the study, whichever occurs first
  Other Names: Single agent Nivolumab

SUMMARY:
The purpose of this study is to determine if nivolumab and ipilimumab are effective treatment for people with pituitary tumors have gotten worse after surgery and radiation.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18
* A pituitary adenoma/carcinoma of any histology

  ° Patients with unresectable tumors that are radiographically (and/or biochemically) consistent with a pituitary adenoma may be considered for enrollment without pathologic confirmation with approval from the principal investigator.
* Progression on imaging following radiotherapy

  ° Patients with pituitary carcinomas in whom there is not felt to be a palliative benefit to treatment with radiotherapy are eligible for enrollment without prior radiotherapy.
* Measurable disease by RANO criteria
* At least 4 weeks have elapsed since the patient last received temozolomide and the patient must have recovered hematologically from other chemotherapeutics
* Karnofsky Performance Status (KPS) greater than or equal to 70
* Screening laboratory values must meet the following criteria:

  * WBC >/= 2000/uL
  * Neutrophils >/= 1500/uL
  * Platelets >/= 100 x 10^3/uL
  * Hemoglobin > 9.0 g/dL
  * AST/ALT </=3 x ULN
  * Total Bilirubin </= 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin <3.0 mg/dL)
* Serum creatinine </= 1.5 x ULN or creatinine clearance (CrCl) >/= 40 mL/min using the Cockcroft-Gault formula
* Women of childbearing potential (WOCBP) must use appropriate method(s) or contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug

  * WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. Women who are not of childbearing potential are not required to use contraception
  * Women of childbearing potential must have a negative serum or urine pregnancy test upon study entry
* Men who are sexually active with women of childbearing potential must use adequate contraception upon study entry until 31 weeks after the last dose of study treatment. Men who are surgically sterile or azoospermic do not require contraception.

Exclusion Criteria:

* A corticosteroid requirement of greater than 4mg per day of dexamethasone (or an equivalent dose). NOTE: Patients requiring a physiologic replacement dose of corticosteroids, who may require stress dose corticosteroids, due to adrenal insufficiency are permitted onto this trial
* Active, known, or suspected autoimmune disease within the past 2 years. NOTE: Subjects are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger
* Patients should be excluded if they have had prior systemic treatment with a CTLA-4 antibody. Prior treatment with PD1 or PD-L1 antibodies are permitted as long as the patient did not experience serious toxicities requiring treatment discontinuation related to prior PD-1 or PD-L1 therapy
* Patients should be excluded if they have a known history of testing positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus antibody (HCV antibody) indicating acute or chronic infection
* Patients should be excluded if they have a known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* History of allergy to study drug components
* History of severe hypersensitivity reaction to any monoclonal antibody
* Women who are pregnant or breast-feeding
* Inability to undergo radiographic surveillance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Radiographic response rate | 36 weeks from baseline
  Radiographic response rate will be assessed by RANO/iRANO

SECONDARY OUTCOMES:
Safety as assessed by CTCAE 5.0 | 36 weeks from baseline
  Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0 will be used to assess safety

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Lin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- [Derived] Dai C, Liang S, Sun B, Kang J. The Progress of Immunotherapy in Refractory Pituitary Adenomas and Pituitary Carcinomas. Front Endocrinol (Lausanne). 2020 Dec 11;11:608422. doi: 10.3389/fendo.2020.608422. eCollection 2020. PMID 33362722
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org